CLINICAL TRIAL: NCT04488341
Title: Effect of Aerobic Exercises on Sex Hormones and Coagulation Factors in Postmenopausal Elderly Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Farid Eid morsy Elsisi, principal investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P.T.REC/012/002676
Record Dates: First submitted 2020-07-14; First posted 2020-07-28 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercises in addition to diet (Other): The study group will receive aerobic exercises in addition to diet recommendations
  Interventions: Other: aerobic exercises in addition to diet recommendations; Other: diet recommendations
- diet recommendations (Other): control group will receive diet recommendations
  Interventions: Other: diet recommendations

INTERVENTIONS:
Other: aerobic exercises in addition to diet recommendations — aerobic exercises time of session 40-50 min initial 10 min warm up exercises on treadmill in low intensity and active phase 20- 30 min intensity will increase until patient reach to target heart rate then intensity decrease until session will be ended by cooling down phase for 10 min . The volunteers will perform exercises 3 times per week for 12 weeks
  Arms: aerobic exercises in addition to diet
Other: diet recommendations — control group will receive diet recommendations for 12 weeks

SUMMARY:
PURPOSE:

to determine the effect of aerobic exercise training on sex hormones and coagulation factors in postmenopausal elderly women

BACKGROUND:

Cardiovascular disease (CVD) is the largest cause of death in women, and the risk of developing CVD increases after menopause . Because thrombosis is thought to be a cause of most acute cardiovascular events, abnormalities in endogenous coagulation and fibrinolysis may play an important role in the risk of an acute cardiovascular event. Aging is also associated with adverse changes in both coagulation and fibrinolysis. For instance, postmenopausal women exhibit higher fibrinogen levels and lower levels of endogenous fibrinolysis. Physical activity and physical fitness have consistently been linked to lower CVD rates in women. In fact, an inverse association between physical activity and total mortality, as well as a 50% reduction in risk of myocardial infarction, has been observed in physically active postmenopausal women. In addition to the numerous other benefits provided by regular physical activity, one of the mechanisms mediating the cardioprotective effect may be changes in the hemostatic system, particularly fibrinolysis

HYPOTHESES:

Aerobic exercises may have no effect on sex hormones and coagulation factors in elderly postmenopausal women

RESEARCH QUESTION:

Do aerobic exercises effect on sex hormones and coagulation factors in elderly postmenopausal women in response to exercises?

DETAILED DESCRIPTION:
It is an interventional study in which 40 women estimated to enroll according to random allocation and assigned into two groups equally. The study group will receive aerobic exercises in addition to diet recommendations while the control group will receive diet recommendations. the aerobic exercises time of session 40-50 min initial 10 min warm up exercises on treadmill in low intensity and active phase 20- 30 min intensity will increase until patient reach to target heart rate then intensity decrease until session will be ended by cooling down phase for 10 min . The volunteers will perform exercises 3 times per week for 12 weeks .coagulation factors(Prothrombin time, Partial Thromboplastin Time , plasminogen activator inhibitor-1 , fibrinogen and tissue plasminogen activator )will be measured and sex hormones (estradiol ,testosterone. sex hormone binding globin ) pre and post intervention

ELIGIBILITY:
Inclusion Criteria:

* • forty Postmenopausal women (60-70 y)

  * Body mass index (BMI) ranged from 35 to 39.9 kg/m2

Exclusion Criteria:

* • regular medications(e.g., β-blockers, α-blockers, digoxin, diuretics, aspirin, nitrates, Presently using hormone replacement therapy (HRT) and non steroidal anti-inflammatory drugs,

  * smoking;
  * cognitive impairment that will make it difficult to partake in the study
  * presence of malignant disease
  * blood donation within the last 6 months
  * Participation as a subject in any type of study or research during the prior 90 days
  * hypertension,
  * having active chronic illness (e.g., rheumatoid arthritis, hyperthyroidism, and inflammatory bowel disease) and diabetes mellitus or other (unstable) endocrine-related diseases
  * personal history of cardiovascular diseases,
  * Orthopedic problems inhibiting exercises.

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
coagulation factors | 12 weeks
  change of selected coagulation factors by blood analysis (plasminogen activator inhibitor-1 ,tissue plasminogen activator ,Prothrombin time ,Partial Thromboplastin time ,fibrinogen )
sex hormones | 12 weeks
  change of (estradiol ,testosterone. sex hormone binding globin )

SECONDARY OUTCOMES:
weight | 12 weeks
  measuring weight in kilograms
height | 12 weeks
  measuring height in meters

CONTACTS AND LOCATIONS:
Overall Officials: hany fm elsisi, phd, Principal Investigator — physical therapy faculty Cairo university
Locations (1):
- Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 2 years after completion study
Access Criteria: journal publishes the study
URL: http://Scholar.cu.edu.eg/p_t